CLINICAL TRIAL: NCT05779540
Title: A New Device to Delay Asphyxiation in Subjects Critically Buried in Avalanche Debris: Efficacy and Pathophysiological Implications
Brief Title: Efficacy and Pathophysiological Implications of a New Asphyxiation Delaying Device
Acronym: SAFEBACK
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Mountain Emergency Medicine (Other)
Collaborators: Medical University Innsbruck (Other); Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Strapazzon, MD PhD, Dr., Institute of Mountain Emergency Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SB1
Record Dates: First submitted 2023-02-13; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Avalanche, Landslide, or Mudslide; Asphyxia; Immersion
Keywords: Avalanche; Avalanche burial; Cardiac arrest; Asphyxia; Emergengy medicine
MeSH Terms: conditions — Asphyxia; Heart Arrest

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Active Device
  Interventions: Device: Safeback SBX
- Control (Sham Comparator): Sham Device
  Interventions: Device: Sham device

INTERVENTIONS:
Device: Safeback SBX — The intervention consists in the test of the active device.
  Arms: Intervention
Device: Sham device — The intervention consists in a similar device to that emits same noise but does not deliver airflow.
  Arms: Control

SUMMARY:
Survival of fully buried avalanche victims depends in major part on a triad of hypoxia, hypercapnia, and hypothermia and therefore decreases rapidly after complete burial. Besides optimizing companion rescue, which still today and even by trained people often takes more than 15 minutes to the extraction of an avalanche victim, prolonging the ability to breath after critical avalanche burial increases survival probability by giving rescuers more time to find and unbury avalanche victims. Based on previous research, the Norwegian company Safeback SE (Bergen, Norway) developed a new non-medical device using an innovative functional principle. The device, called the Safeback SBX (Safeback SE, Bergen, Norway), should make it possible to prevent asphyxia by delivering fresh air to the air pocket. Company claims to achieve a prolongation of survival up to over 60 minutes, giving companion rescuers as well as professional rescue teams more time to get access to the victim. Technical tests conducted by the developing company already provided some promising results regarding the general functioning. However, this study is needed to provide the scientific evidence of the effectiveness and influence on physiologic parameters buried in snow debris humans under realistic conditions.

ELIGIBILITY:
Inclusion Criteria:

- healthy ASA I subjects

Exclusion Criteria:

* ASA class II or higher
* chronic high degree cardiovascular or pulmonary disease
* claustrophobia
* psychiatric or neurological disease
* long-term medication
* pregnant woman
* no informed consent
* history of fever or serious cough in the past two weeks
* current Covid-19 symptoms or recently tested positive for Covid-19
* body temperature ≥ 37.5°on test days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Time limit | From baseline up to 60 minutes
  Reaching a predefined time limit (min)
Physiological threshold | From baseline up to 60 minutes
  Time to reach a SpO2 threshold up to <75% (min)

SECONDARY OUTCOMES:
End-tidal CO2 (EtCO2) | Changes from baseline (measurement at 0 min) -> snow-breathing phase (5min, 15min, and timepoint immediately before interruption [up to 60 min) (countinuous monitoring)
  Changes in EtCO2 (mmHg)
Minute ventilation (VE) | Changes from baseline (measurement at 0 min) -> snow-breathing phase (5min, 15min, and timepoint immediately before interruption [up to 60 min) (countinuous monitoring)
  Changes in VE (L/min)
Cerebral Regional Oxygen Saturation (rSO2) | Changes from baseline (measurement at 0 min) -> snow-breathing phase (5min, 15min, and timepoint immediately before interruption [up to 60 min) (countinuous monitoring)
  Changes in rSO2 (%)
NASA-task load index (NASA-TLX) questionnaire (perceived workload) | Change from basal measurement (before hypoxia exposure) to post-exposure measurement (after hypoxia exposure - up to 60 min)
  Changes in NASA-task load index (NASA-TLX) questionnaire (numerical scale)
Reactive oxygen species - ROS | Change from basal measurement (before hypoxia exposure) to post-exposure measurement (after hypoxia exposure - up to 60 min)
  Changes in ROS in saliva samples (μmol/min)
Total antioxidant capacity - TAC | Change from basal measurement (before hypoxia exposure) to post-exposure measurement (after hypoxia exposure - up to 60 min)
  Changes in TAC in saliva samples (mM)

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Strapazzon, Dr., Principal Investigator — Institute of Mountain Emergency Medicine, Eurac Research
Locations (1):
- Institute of Mountain Emergency Medicine, Eurac Research, Bolzano, Bz, Italy

REFERENCES:
- [Background] Falk M, Brugger H, Adler-Kastner L. Avalanche survival chances. Nature. 1994 Mar 3;368(6466):21. doi: 10.1038/368021a0. No abstract available. PMID 7969398
- [Background] Wik L, Brattebo G, Osteras O, Assmus J, Irusta U, Aramendi E, Mydske S, Skaalhegg T, Skaiaa SC, Thomassen O. Physiological effects of providing supplemental air for avalanche victims. A randomised trial. Resuscitation. 2022 Mar;172:38-46. doi: 10.1016/j.resuscitation.2022.01.007. Epub 2022 Jan 19. PMID 35063621
- [Background] Strapazzon G, Paal P, Schweizer J, Falk M, Reuter B, Schenk K, Gatterer H, Grasegger K, Dal Cappello T, Malacrida S, Riess L, Brugger H. Effects of snow properties on humans breathing into an artificial air pocket - an experimental field study. Sci Rep. 2017 Dec 15;7(1):17675. doi: 10.1038/s41598-017-17960-4. PMID 29247235
- [Derived] Eisendle F, Roveri G, Rauch S, Thomassen O, Dal Cappello T, Assmus J, Malacrida S, Kammerer T, Schweizer J, Borasio N, Dorck V, Falk M, Falla M, Fruzzetti N, Maxenti M, Mydske S, Sasso GM, Vinetti G, Wallner B, Brattebo G, Brugger H, Strapazzon G. Respiratory Gas Shifts to Delay Asphyxiation in Critical Avalanche Burial: A Randomized Clinical Trial. JAMA. 2025 Oct 8;334(19):1720-7. doi: 10.1001/jama.2025.16837. Online ahead of print. PMID 41060661